CLINICAL TRIAL: NCT06710626
Title: CONVOY: An Early Feasibility Study of Neural Control of Assistive Devices Via Brain-Computer Interface Technology
Brief Title: Control of Assistive Devices Via Brain-Computer Interface Technology
Acronym: CONVOY
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Neuralink Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N1-EFS-100
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Tetraplegia/Tetraparesis; Amyotrophic Lateral Sclerosis (ALS); Quadriplegia; Spinal Cord Injury (SCI); Spinal Cord Injury Cervical
Keywords: brain computer interface; robotic arm; assistive device; Neuralink N1 Implant; Neuralink; N1 Implant; ALS; Spinal cord injury; Quadriplegia; tetraplegia; Robot; external device control; neuroprosthetics
MeSH Terms: conditions — Quadriplegia; Amyotrophic Lateral Sclerosis; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: The study is a prospective, longitudinal, non-randomized, open-label, single-arm early feasibility study (EFS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single (Other)
  Interventions: Device: Assistive Robotic Arm

INTERVENTIONS:
Device: Assistive Robotic Arm — The intervention involves using the N1 Implant, a wireless brain-computer interface (BCI), to enable participants to control the Assistive Robotic Arm through neural signals.
  Other Names: BCI controlled robotic arm

SUMMARY:
The CONVOY Study is a clinical trial designed to explore the feasibility of participants from the PRIME Study (NCT06429735) using the N1 Implant to control various assistive devices. The main goal is to determine whether participants can successfully modulate their brain activity to control devices, such as an Assistive Robotic Arm (ARA). This study will assess the effectiveness, consistency, and safety of neural control using the ARA and other assistive devices.

ELIGIBILITY:
Inclusion Criteria:

* Continued enrollment in the PRIME Study.
* Implanted with the N1 Implant.

Exclusion Criteria:

* Explantation or deactivation of the N1 Implant.
* Insufficient N1 Implant BCI performance demonstrated.
* Lack of a suitable physical space to perform research sessions.
* Any condition which, in the opinion of the Investigator, would compromise the candidate's ability to safely participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2031-05-25 (Estimated); Study Completion 2031-05-25 (Estimated)

PRIMARY OUTCOMES:
Ability of participants to modulate brain activity for controlling an assistive device via the N1 Implant. | 3-months following first use of the assistive device

SECONDARY OUTCOMES:
Rate of Device-Related Adverse Events (AE) | Up to 72 months after enrollment
Assessment of Quality of Life Using the Psychosocial Impact of Assistive Devices Scale (PIADS) | From enrollment, every 3 months, up to 72 months
Change in Assistive Technology Device Predisposition Assessment (ATD PA) Score | From enrollment, every 3 months, up to 72 months

CONTACTS AND LOCATIONS:
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Neuralink Website — https://neuralink.com/